CLINICAL TRIAL: NCT00003908
Title: Evaluation of the Combination of Docetaxel (Taxotere)/ Carboplatin in Patients With Metastatic or Recurrent Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: S9902 Docetaxel Plus Carboplatin in Treating Patients With Metastatic or Recurrent Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067086; S9902 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-05-21 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Head and Neck Cancer
Keywords: recurrent metastatic squamous neck cancer with occult primary; metastatic squamous neck cancer with occult primary squamous cell carcinoma; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: carboplatin
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of docetaxel plus carboplatin in treating patients who have metastatic or recurrent head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the survival of patients with metastatic or recurrent squamous cell carcinoma of the head and neck receiving docetaxel and carboplatin. II. Assess time to treatment failure and response rate (unconfirmed and confirmed complete and partial response) in this patient population. III. Evaluate the toxicities of this regimen in this patient population.

OUTLINE: Patients receive docetaxel IV over 1 hour immediately followed by carboplatin IV over 30 minutes on day 1. Courses repeat every 3 weeks in the absence of unacceptable toxicity or disease progression. Patients are followed every 3 months for 1 year, every 6 months for 2 years, then annually thereafter until death.

PROJECTED ACCRUAL: A total of 62 patients will be accrued for this study over 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven squamous cell carcinoma of the head and neck Metastatic disease at diagnosis OR Persistent, metastatic or recurrent disease following surgery and/or radiotherapy No newly diagnosed nonmetastatic disease Bidimensionally measurable disease Demonstrated progressive disease if only measurable site is within a previous radiotherapy port

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: SWOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 OR Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2 times upper limit of normal (ULN) SGOT or SGPT no greater than 1.5 times ULN Alkaline phosphatase no greater than 2.5 times ULN Renal: Calcium no greater than upper limit of normal (ULN) Creatinine no greater than 1.5 times ULN OR Creatinine clearance at least 60 mL/min Other: Not pregnant or nursing Fertile patients must use effective contraception No other prior malignancy within the past 5 years except adequately treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or any adequately treated stage I or II cancer that is currently in complete remission No neuropathy sensory greater than grade 1 No history of hypersensitivity reaction to Polysorbate 80

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent biologic therapy Chemotherapy: No prior carboplatin or cisplatin No prior chemotherapy for recurrent disease No other concurrent chemotherapy Endocrine therapy: No concurrent hormonal therapy (except oral contraceptives or treatment for osteoporosis) Radiotherapy: See Disease Characteristics At least 28 days since prior radiotherapy and recovered No concurrent radiotherapy Surgery: See Disease Characteristics At least 28 days since prior surgery and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 1999-11; Primary Completion 2004-06 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Weekly while on protocol treatment, then every 3 months for 1 year, then every 6 months for 2 years.
  Overall survival was defined as the duration from the date of registration to the date of death due to any cause. Patients last known to be alive were censored at the date of last contact.

SECONDARY OUTCOMES:
Progression-Free Survival | Every 6 weeks until progression of disease.
  Progression-Free Survival was defined as the duration between the date of registration and the date of first documentation of progression of disease or death due to any cause. Progression of disease was defined as a 50% increase in the sum of products of perpendicular diameters of measurable lesions or an increase of at least 10 square centimeters, whichever was smaller, or clear worsening of non-measurable lesions in the opinion of the treating investigator, appearance of new lesions, reappearance of lesions that had previously disappeared, or symptomatic deterioration.
Response | Every 6 weeks while on protocol treatment.
  Response was defined as a confirmed or unconfirmed complete or partial response. A complete response (CR) was defined as disappearance of all disease. A partial response (PR) was defined as a 50% decrease or greater in the sum of perpendicular diameters of all measurable lesions. A CR or PR was defined as confirmed if there were two consecutive determinations at least 3 weeks apart.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfram E. Samlowski, MD, BA, Study Chair — University of Utah
Locations (85):
- United States (85):
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Cancer Services, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- [Result] Samlowski WE, Moon J, Kuebler JP, Nichols CR, Gandara DR, Ozer H, Williamson SK, Atkins JN, Schuller DE, Ensley JF. Evaluation of the combination of docetaxel/carboplatin in patients with metastatic or recurrent squamous cell carcinoma of the head and neck (SCCHN): a Southwest Oncology Group Phase II study. Cancer Invest. 2007 Apr-May;25(3):182-8. doi: 10.1080/07357900701209061. PMID 17530488